CLINICAL TRIAL: NCT04940611
Title: SPOTLITE: Prospective Observational Study on the Clinical Outcomes of Surgical Interventions in Complex Fistulizing Conditions (CPF-CD, CD-RVF, CCF)
Brief Title: A Study of Surgical Interventions in Fistulizing Conditions
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alofisel-5007
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Crohns Disease; Fistula; Rectovaginal Fistula; Complex Perianal Fistula; Complex Cryptoglandular Fistula
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Fistula; Rectovaginal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants With CPF-CD: Participants diagnosed with CPF-CD will undergo surgical intervention according to their clinic's standard practice to treat the index fistula, and will be observed prospectively for 24 months post-index surgery.
- Participants With CD-RVF: Participants diagnosed with CD-RVF will undergo surgical intervention according to their clinic's standard practice to treat the index fistula, and will be observed prospectively for 24 months post-index surgery.
- Participants With CCF: Participants diagnosed with CCF will undergo surgical intervention according to their clinic's standard practice to treat the index fistula, and will be observed prospectively for 24 months post-index surgery.

SUMMARY:
In this study, participants with complex fistulizing conditions will be treated with surgical interventions according to their clinic's standard practice.

The aim of the study is to generate real-world evidence on standard of care for surgical interventions and related outcomes when treating complex fistulizing conditions.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with complex fistulizing conditions (CPF-CD, CD develops CD-RVF and CCF) who are currently undergoing surgical intervention in the real world clinical setting.

The study will enroll approximately 750 participants. The data will be collected prospectively at the study sites and will be recorded into electronic data capture forms (EDCs). Participants will be enrolled to the following observational cohorts:

* Participants With CPF-CD
* Participants With CD-RVF
* Participants With CCF

This multi-center study will be conducted in the United States, Canada, Europe, and Israel. Participants undergoing surgical interventions to treat fistulas will be enrolled from surgical and gastrointestinal (GI) specialty sites. The overall duration of the study will be 24 months. Data will be collected at baseline with follow-up information collected approximately every 3 to 6 months.

ELIGIBILITY:
Inclusion Criteria:

Participants with CPF-CD

1. CPF-CD that meets one or more of the following criteria:

   * High inter-sphincteric, high trans-sphincteric, extra-sphincteric or supra-sphincteric fistula, or
   * Presence of greater than or equal to (>=) 2 external openings, or
   * Associated perianal abscess(es)
2. Physician has made the decision to treat with a specific surgical intervention. Procedures may include:

   * Fistulotomy, fistula plug, fibrin glue, advancement flap (AF), ligation of inter-sphincteric fistula tract (LIFT), flap repair, fistulectomy, proctectomy, stem cell therapy, other; and seton for palliative purposes.

Participants with CD-RVF: Rectovaginal fistula per physician diagnosis

1. Physician has made the decision to treat with a specific surgical intervention. Procedures may include:

* Fistulotomy, fistula plug, fibrin glue, AF, LIFT, flap repair, fistulectomy, proctectomy, stem cell therapy, gracilis muscle interposition/tissue grafts, martius procedure, abdominal procedures, other; and seton use for palliative purposes.

Participants with CCF:

1. Complex cryptoglandular fistula that meets one or more of the following criteria:

   * Mid or high trans-sphincteric, or
   * Anterior in women, or
   * Horseshoe fistula
2. Physician has made the decision to treat with a specific surgical intervention. Procedures may include:

   * Fistulotomy, fistula plug, fibrin glue, AF, LIFT, flap repair, fistulectomy, proctectomy, stem cell therapy, other; and seton use for palliative purposes

Exclusion Criteria:

Participants who meet any below mentioned criterion among CPF-CD, CD-RVF, and CCF diagnosis will be excluded from the study.

1. Current participation in interventional clinical trials.
2. Has CPF-CD: fistula connection to bladder or another organ
3. Has CCF: diagnosis of Inflammatory Bowel Disease (IBD), including Ulcerative Colitis, and Crohn's Disease (CD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing surgical interventions to treat fistulas (CPF-CD, CD-RVF and CCF) from surgical and GI specialty sites.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Clinical Remission of Fistula | Baseline up to 24 months
  Clinical remission for Complex perianal fistula in Crohn's Disease (CPF-CD) and Complex Cryptoglandular Fistula (CCF) is defined as closure of all index treated external fistula openings that were draining at baseline as assessed clinically despite gentle finger compression. Clinical remission for Rectovaginal fistula with Crohn's Disease (CD-RVF) is defined as epithelization of the index external fistula opening (vaginal opening) compared to baseline.

SECONDARY OUTCOMES:
Percentage of Participants With Post-surgical Complications | Baseline, 3, 6, 12 and 24 months post-index surgery
  Post-surgical complications for CPF-CD and CCF is defined as post-index surgery perianal pain, bleeding, infection, urinary retention, delayed or poor wound healing, anal stenosis, and fecal incontinence related to index surgery. Post-surgical complications for CD-RVF is defined as post-index surgery vaginal bleeding, infection, urinary retention, urinary tract infections (UTIs), discharge, delayed or poor wound healing, anal stenosis, fecal incontinence, and pain with intercourse or others related to index surgery.
Percentage of Participants who Achieve Combined Remission | Baseline, 3, 6, 12 and 24 months post-index surgery
  Combined remission for CPF-CD and CCF is defined as closure of all index external fistula openings treated with surgery that were draining at baseline as assessed clinically despite gentle finger compression, and absence of fluid collections greater than (>) 2 centimeter (cm) in at least 2 dimensions, as confirmed by pelvic magnetic resonance imaging (MRI) or other imaging procedure. Combined remission for CD-RVF is defined as 100 percent (%) cessation of drainage on both clinical exam with deep palpation (deeper bimanual exam/palpation with speculum and/or anoscope) and epithelization of the index external fistula opening (vaginal opening) compared to baseline; and absence of fluid collection as assessed by MRI or other imaging procedure.
Percentage of Participants who Achieve Cessation of Drainage in Treated Fistula | Baseline, 3, 6, 12 and 24 months post-index surgery
  Cessation of drainage for CPF-CD and CCF is defined as 100% cessation of drainage from index treated fistula, as assessed clinically. Cessation of drainage for CD-RVF is defined as 100% cessation of drainage on clinical exam with deep palpation (deeper bimanual exam/palpation with speculum and/or anoscope) from the index treated fistula.
Percentage of Participants With Relapse of Fistula in Clinical Remission | Baseline, 3, 6, 12 and 24 months post-index surgery
  Relapse for CPF-CD and CCF is defined as reopening of any surgically treated index fistulae as clinically assessed; or the development of a perianal fluid collection >2 cm in at least 2 dimensions of the perianal fistula(s) treated, confirmed by MRI assessment or other imaging procedure; or drainage. Relapse for CD-RVF is defined as reopening of any surgically treated index fistulae as clinically assessed; or appearance of fluid collection as assessed by MRI or other imaging procedure; or drainage.
Percentage of Participants With New Perianal Abscess | Baseline, 3, 6, 12 and 24 months post-index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- United States (13):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of South Florida - PARENT, Tampa, Florida
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - GI Alliance - Baton Rouge, Baton Rouge, Louisiana
  - Lenox Hill Hospital PRIME, New York, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Premier Health, Dayton, Ohio
  - Penn Medicine PA, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center- GI Endoscopy Lab, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Colon & Rectal Clinic, Houston, Texas
- AKH - Medizinische Universitat Wien, Vienna, Austria
- Belgium (5):
  - UZ Antwerpen, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Jessa Ziekenhuis Hospital, Hasselt
  - Clinique CHC MontLegia, Liège
  - AZ Delta, Roeselare
- St. Pauls Hospital, Vancouver, British Columbia, Canada
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - NH Hospital a.s.Nemocnice Horovice, Hořovice
  - Fakultni nemocnice Olomouc, Olomouc
- France (7):
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Bouches-du-Rhone
  - Fondation Maison Sante Bagatelle, Talence, Gironde
  - CHU de Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - CHRU Hopital Claude Huriez, Lille, Nord
  - CHU de Rouen - Hopital Charles Nicolle, Rouen, Seine Maritime
  - Groupe Hospitalier Diaconesses - Hopital De La Croix Saint Simon, Paris
  - Hopital Saint Joseph - Paris, Paris
- Israel (4):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Rambam Health Care Center, Haifa
  - Wolfson Medical Center, Holon
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Istituto Clinico Humanitas, Rozzano, Milano, Italy
- Netherlands (2):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - UMC Utrecht, Utrecht
- United Kingdom (3):
  - Broomfield Hospital, Chelmsford, Essex
  - Nottingham University Hospital, Nottingham, Nottinghamshire
  - Royal Victoria Infirmary., Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/60acd8531f1122001e30a7ff?idFilter=%5B%22Alofisel-5007%22%5D